CLINICAL TRIAL: NCT03936608
Title: Electrocardiogram for Programming in Cardiac Resynchronization Therapy
Brief Title: ECG for Programming in CRT
Acronym: EPIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left Washington University
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201901208
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Systolic Heart Failure; Cardiac Resynchronization Therapy; Electrocardiography
Keywords: CRT Programming
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Individualized RV-LV Pacing Offset (Experimental)
  Interventions: Device: Programming individualized RV-LV pacing offset to optimize ECG
- No RV-LV Pacing Offset (Active Comparator)
  Interventions: Device: Nominally programming CRT device without RV-LV offset

INTERVENTIONS:
Device: Programming individualized RV-LV pacing offset to optimize ECG — After CRT device implant, participants will undergo physiologic evaluations at various (up to 10 or more) RV-LV offset settings including ECGs. The RV-LV offset that optimizes the paced QRS morphology on ECG will be programmed.
  Arms: Individualized RV-LV Pacing Offset
Device: Nominally programming CRT device without RV-LV offset — After CRT device implant, participants will undergo physiologic evaluations at various (up to 10 or more) RV-LV offset settings including ECGs. Nominal standard-of-care CRT programming with no RV-LV offset will be programmed.
  Arms: No RV-LV Pacing Offset

SUMMARY:
Patients with heart failure and left bundle branch block benefit from Cardiac Resynchronization Therapy (CRT) that delivers pacing from right ventricle (RV) and left ventricle (LV) synchronously, resulting in electrical ventricular resynchrony followed by revere structural cardiac remodeling and thereby reduced heart failure symptoms, hospitalizations and death. It is not known if programming an individually optimized RV-LV pacing offset to maximize electrical resynchrony can improve benefit from CRT.

The proposed study is a randomized controlled trial in patients undergoing implant of a CRT pacemaker/defibrillator device for clinical indications to evaluate benefit of RV-LV offset programming using electrocardiogram (ECG) vs. standard nominal CRT programming without RV-LV offset. Patients receiving CRT devices will be randomized to either (A) active intervention of programming RV-LV pacing offset to optimize ECG or to (B) active control of nominally programming CRT device without RV- LV offset. The patients will be followed to evaluate change in echocardiogram, quality of life, functional evaluation and a blood marker for heart failure.

DETAILED DESCRIPTION:
Once the eligibility for the study is determined and patient has consented for participation, all study participants will undergo a baseline evaluation (within 6 weeks prior to 2 weeks after CRT device implant/upgrade). Echocardiogram, quality-of-life questionnaire, 6-minute hall walk, blood test, vital signs, ECGs, device interrogation and baseline demographic and medical history including chart review will be obtained. After CRT device implant/upgrade, participants will undergo physiologic evaluations at various (up to 10 or more) RV-LV offset settings including ECGs and echocardiography. A randomized assignment using a random allocation table in REDCap will be used to program patients to (A) intervention or (B) control RV-LV offset setting. Patients will return for study follow-up between 3-12 months. Follow-up evaluations will include echocardiography, quality-of-life questionnaire, 6-minute hall walk test, blood test, vital signs, ECGs, device interrogation, and follow-up medical history including chart review. The patients will continue to be in extended follow-up through review of their medical charts till the end of the study (12 months from date of CRT implant/upgrade of the the last study participant).

Treatment and control arms: All study patients will receive standard of care clinically indicated medical and device therapy per their treating physicians. After implant of a clinically indicated CRT device or upgrade of a preexisting pacemaker or defibrillator device to CRT system, participants will be randomized 1:1 to treatment arms (A) active intervention of programming individualized RV-LV pacing offset to optimize ECG or to (B) active control of nominally programming CRT device without RV-LV offset. Of note, both intervention and control treatment are active FDA-approved CRT therapies and no investigational device or programming will be used, and no clinically indicated treatment will be withheld from any patient. At any time, if in the judgment of the patient's treating physicians or the research team, any treatment including CRT programming different from the study protocol is necessitated for clinical reasons, the appropriate clinically indicated changes will be made. At the end of the study, if the participant is clinically doing well and the programmed CRT settings are deemed clinically appropriate they will be retained, else the CRT programming may be changed as per standard of care.

Enrolled participants who have a failed or unsatisfactory LV lead implant will not be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age who are able to give consent.
* Diagnosis of systolic heart failure.
* Planned to undergo new CRT device implant (or upgrade of preexisting pacemaker or defibrillator device to CRT system) for standard clinical indications.
* Expected to have over 95% heart beats resynchronized with CRT (absence of competing arrhythmias or plans to not immediately activate CRT therapy).

Exclusion Criteria:

* Unable to comply with the study follow-up.
* Life expectancy ≤1 year.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Noheria, MBBS, SM, Principal Investigator — Washington University School of Medicine; Sandeep Sodhi, MD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individualized RV-LV Pacing Offset | No RV-LV Pacing Offset
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individualized RV-LV Pacing Offset | No RV-LV Pacing Offset | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 66 [50 to 82] | 43 [33 to 53] | 54.5 [33 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Randomization Groups [Count of Participants; unit: Participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is Echocardiographic LV End-systolic Volume.
Description: LV end-systolic volume is a reliable surrogate for clinical outcomes in clinical heart failure trials.
Time Frame: 3-12 months
Population: Study prematurely terminated, no data analysis was performed
Arm/Group | Individualized RV-LV Pacing Offset | No RV-LV Pacing Offset
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Individualized RV-LV Pacing Offset | No RV-LV Pacing Offset
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT03936608/Prot_SAP_001.pdf